CLINICAL TRIAL: NCT01103856
Title: Test of an Intervention to Improve HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas Giordano, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH085527-01A1 (NIH); 1R01MH085527-01A1 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: HIV Infection
Keywords: HIV; adherence to care; retention in care; patient navigation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Mentor Intervention (Experimental): The patient mentor intervention from TSHC has been adapted to the inpatient setting. Participants randomized to that arm will receive 2 sessions with a patient mentor during their hospitalization, as well as 5 phone call sessions over the 10 weeks after discharge and a brief meeting between the subject and the mentor when the subject attends their first outpatient visit at TSHC after discharge.
  Interventions: Behavioral: Patient Mentor Intervention
- HIV transmission risk reduction (Placebo Comparator): Participants randomized to the control arm will receive an attention control intervention delivered by a patient educator who is not an HIV patient mentor. We will use a modified version of the RESPECT intervention for our attention control group. Similar to the active intervention, these patients will receive 2 sessions in the hospital and 5 phone calls over 10 weeks after discharge.
  Interventions: Behavioral: HIV transmission risk reduction

INTERVENTIONS:
Behavioral: Patient Mentor Intervention — The first session includes an exploration of needs, barriers, and facilitators to HIV care. HIV educational materials are introduced to identify areas of need. Mentors will address concerns and possible barriers to care using their own experiences. Mentors will encourage participants to set goals related to acquisition of care following discharge and how to address possible barriers to that goal. The second session will reinforce the first session. Mentors will call the patient 5 times over the 10 weeks after discharge. These phone calls will be brief and goal centered, to either reinforce positive behavior if the patient is in care, or continue to help the patient re-engage in outpatient HIV care.
  Other Names: MAPPS; Mentor Approach for Promoting Patient Self-care
  Arms: Patient Mentor Intervention
Behavioral: HIV transmission risk reduction — The control intervention is a modification of the project RESPECT intervention. We will use material from sessions 1, 2, and 3 of the RESPECT enhanced counseling intervention. These interactions will include a personalized assessment of risk behaviors and changing condom use self-efficacy. The second interaction will build on material covered during the first interaction, with additional focus on condom use attitudes. The counselors will call the patient 5 times in the 10 weeks after discharge. These phone-based sessions will be brief and goal centered, to reinforce safe HIV transmission behaviors.
  Other Names: RESPECT
  Arms: HIV transmission risk reduction

SUMMARY:
At Thomas Street Health Center (TSHC), one of the largest outpatient HIV clinics in the country, we developed a structured, theory-based, Patient Mentor Program to improve retention in HIV primary care. Many patients with HIV infection hospitalized at Ben Taub General Hospital (BTGH) do not successfully return to TSHC after discharge from the hospital. The purpose of this study is to test the efficacy of a patient mentor intervention in a 5-year randomized, controlled trial in more than 430 socio-economically and racially diverse HIV-infected patients hospitalized at BTGH. We hypothesize that the intervention will meaningfully increase retention in HIV primary care after discharge compared to an attention control.

ELIGIBILITY:
Inclusion Criteria:

1) Hospitalized at BTGH; 2) expected to be in the hospital for at least one more night at the time of enrollment; 3) at least 18 years of age at enrollment; 4) able to speak English or Spanish; 5) HIV infected, whether previously diagnosed or diagnosed this hospital stay; 6) cognitively aware enough to provide informed consent and participate in the study. Patients who are temporarily cognitively incapacitated (e.g., from an acute process) will be followed and approached for enrollment if and when they are cognitively and physically capable of participating in the study.

Exclusion Criteria:

1) Intending to use a source of HIV primary care other than TSHC after discharge from the hospital, because TSHC-specific mentoring is not relevant to them and the data on their appointments after discharge cannot be tracked; 2) in the opinion of the primary medical team, likely to be discharged to an institutional setting; 3) in the opinion of the primary medical team caring for the patient, likely to die in the hospital or be discharged to hospice; 4) cognitive impairment that in the opinion of the primary medical team caring for the patient is not expected to improve by discharge; 5) prisoner at admission and expected to be discharged back to prison or jail; 6) having had an HIV primary care visit in at least 3 of the 4 previous quarter-years AND having had at least 3 consecutive HIV VL<400 c/mL over at least 6 months, the most recent of which is within 3 months of enrollment; 7) enrolled in any other research project with prospective follow-up; 8) already enrolled in this study at any time.

For the purposes of this study, "prisoner" will be defined in accordance with Federal regulations, as "any individual involuntarily confined or detained in a penal institution...[including] individuals sentenced to such an institution under a criminal or civil statute, individuals detained in other facilities by virtue of statutes or commitment procedures which provide alternatives to criminal prosecution or incarceration in a penal institution, and individuals detained pending arraignment, trial, or sentencing…Parolees who are detained in a treatment center as a condition of parole are prisoners; however, persons living in the community and sentenced to community-supervised monitoring, including parolees, are not prisoners." Parolees meeting the definition of prisoner will be ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2010-05; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Engaged in outpatient HIV care | 6 Months
  A composite of attending at least one HIV primary care visit within 30 days of discharge AND at least one between 31 and 180 days AND, for patient with an indication for ART, achieving a one log10 decrease in HIV VL or maintaining a VL <400 c/mL at 180 days after discharge.

SECONDARY OUTCOMES:
Completion of at least one HIV primary care visit at TSHC within 30 days of discharge, health services use, changes in CD4 cell count and HIV VL, and quality of life. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Giordano, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Giordano TP, Cully J, Amico KR, Davila JA, Kallen MA, Hartman C, Wear J, Buscher A, Stanley M. A Randomized Trial to Test a Peer Mentor Intervention to Improve Outcomes in Persons Hospitalized With HIV Infection. Clin Infect Dis. 2016 Sep 1;63(5):678-686. doi: 10.1093/cid/ciw322. Epub 2016 May 23. PMID 27217266